CLINICAL TRIAL: NCT06175143
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase Ib Clinical Trial to Evaluate the Tolerability, Safety, Pharmacokinetics, Immunogenicity, and Preliminary Efficacy of GR2002 Injection in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety and Efficacy of GR2002 Injection in Patients With Atopic Dermatitis.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR2002-002
Record Dates: First submitted 2023-11-23; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Atopic Dermatitis
Keywords: TSLP
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GR2002 injection 1 (Experimental): GR2002 injection dose 1/Placebo，multiple-dose，Subcutaneous，high frequency
  Interventions: Biological: GR2002 injection
- GR2002 injection 2 (Experimental): GR2002 injection dose 2/Placebo，multiple-dose，Subcutaneous，high frequency
  Interventions: Biological: GR2002 injection
- GR2002 injection 3 (Experimental): GR2002 injection dose 3/Placebo，multiple-dose，Subcutaneous，high frequency
  Interventions: Biological: GR2002 injection
- GR2002 injection 4 (Experimental): GR2002 injection dose 3/Placebo，multiple-dose，Subcutaneous，low frequency
  Interventions: Biological: GR2002 injection

INTERVENTIONS:
Biological: GR2002 injection — TSLP monoclonal antibody

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase Ib clinical trial evaluating the safety tolerability, pharmacokinetics, immunogenicity and preliminary efficacy of GR2002 Injection in patients with moderate to severe atopic dermatitis. The dosing period was 12 weeks and followed up to 20 weeks.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patients need to meet Williams diagnostic criteria, have had AD for at least 1 year, and:EASI ≥16, IGA score ≥3, and AD involvement of ≥10% of BSA;
2. Inadequate response or intolerance to prior topical glucocorticoid (TCS) therapy for the treatment of AD;
3. Voluntary informed consent.

Main Exclusion Criteria:

1. Current malignancy or history of malignancy;
2. History of vital organ transplantation or hematopoietic stem cell/bone marrow transplantation;
3. Subjects may have active Mycobacterium tuberculosis infection;
4. Systemic anti-infective therapy required for chronic or acute active infection within 4 weeks prior to the baseline visit;
5. History of known or suspected immunosuppression;
6. Presence of skin comorbidities that may interfere with evaluation;
7. Suspected or confirmed allergy to the test drug (including excipients, similar drugs);
8. History of alcohol or drug abuse within 3 months prior to screening；
9. Pregnant or lactating women who need to breastfeed；
10. Major surgery planned during the trial；
11. The elution cycle of the drug of interest is not met at the baseline；
12. Subjects of childbearing potential and partners refusing to use highly effective contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Within 20 weeks
  Incidence of AEs.

SECONDARY OUTCOMES:
Pharmacokinetics parameters | Within 20 weeks
  concentration of GR2002
IGA Response | Within 20 weeks
  Proportion of subjects with an IGA score of 0-1 and a decrease of ≥2 points from baseline
EASI 50/75/90 Response | Within 20 weeks
  Proportion of subjects with ≥50%, ≥75%, and ≥90% improvement in EASI score
Percentage change in BSA score | Within 20 weeks
  Percentage change from baseline in BSA involvement in atopic dermatitis lesions
Proportion of Subjects With Weekly Mean Reduction in Daily Peak Pruritus NRS of ≥4/≥3 | Within 20 weeks
  Proportion of subjects with ≥4/3-point decrease in PP-NRS from baseline
immunogenicity | Within 20 weeks
  Detection of anti-drug antibody(ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, PHD, Principal Investigator — Peking University People's Hospital; Cheng Zhou, PHD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China